CLINICAL TRIAL: NCT04597749
Title: Nebula Study: Comparison of Sleep Screener Apps and Home Sleep Apnea Tests to Polysomnography
Brief Title: Nebula Study - Screener Apps and HSAT vs. PSG Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SLP-20-06-01
Record Dates: First submitted 2020-08-31; First posted 2020-10-22 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Sleep Apnea, Obstructive
Keywords: OSA; Sleep Apnea; OSA Screeners; Home Sleep Apnea Test
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Concurrent PSG, HSAT, and Screener App Test (Experimental): Participants will undergo a single night baseline PSG test with concurrent HSAT tests as well as non-contact screening mobile apps through a smartphone.
  Interventions: Diagnostic Test: PSG; Diagnostic Test: Home Sleep Apnea Test with FDA cleared devices; Other: Non-Contact Screening App

INTERVENTIONS:
Diagnostic Test: PSG — In-lab sleep polysomnography test
Diagnostic Test: Home Sleep Apnea Test with FDA cleared devices — In-lab HST test
Other: Non-Contact Screening App — Non-Contact Sleep Apnea Screening Applications at bedside table to assess for sleep apnea.

SUMMARY:
This is a prospective, unblinded, open-label, single group study. All subjects will undergo concurrent screener app, HSAT testing, and in-lab polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 years of age or older
* Participant is willing to provide informed consent
* Participant is willing to participate in all study related procedures

Exclusion Criteria:

* Unable to cease PAP therapy during PSG (if currently using)
* Requires use of oxygen therapy during sleep
* Diagnosis of untreated clinically relevant sleep disorder (other than SDB)
* Pregnant
* Participant is unsuitable to participate in the study in the opinion of the investigator
* Participant has a permanent pacemaker, sustained non-sinus cardiac arrhythmias, and/or takes alpha blocker or short acting nitrate medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
AHI value. Clinical decision for treatment output (Y to CPAP or N to CPAP) of Screener apps and HSAT compared to PSG. | Day 1
  The PSG clinical decision for treatment is defined as AHI≥15. Screener apps and HSATs provide AHI values that will be used for comparison.

SECONDARY OUTCOMES:
OSA severity categories (normal, mild, moderate, severe) of Screnner apps and HSAT compared to PSG. | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Clayton Sleep Institute, Maplewood, Missouri, United States

IPD SHARING:
Plan to Share IPD: No